CLINICAL TRIAL: NCT05742243
Title: Abatacept Combined With Nasal Insulin to Preserve Beta-cell Function in Recently-diagnosed Type 1 Diabetes
Brief Title: Insulin and Abatacept in Recently-diagnosed Type 1 Diabetes
Acronym: IAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.079
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus, Type 1
Keywords: Abatacept; Nasal insulin; Beta-cell function; Glucose intolerance; Immune responses; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Intolerance; Hypoglycemia | interventions — Abatacept; Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abatacept and nasal insulin (Active Comparator): Abatacept (CTLA4-Ig; 50 mg for participant weight <25 kg, 87.5 mg for participant weight 25-50 kg, 125 mg for participant weight >50 kg) will be injected subcutaneously once per week and nasal insulin (Humulin R®, 100 Units/mL) will be inhaled for 10 consecutive days initially and twice per week thereafter, for 48-weeks.
  Interventions: Drug: Abatacept (CTLA4-Ig) and nasal insulin (Humulin R®)
- Abatacept and nasal placebo (Placebo Comparator): Abatacept (CTLA4-Ig; 50 mg for participant weight <25 kg, 87.5 mg for participant weight 25-50 kg, 125 mg for participant weight >50 kg) will be injected subcutaneously once per week and nasal placebo (0.9% sodium chloride) will be inhaled for 10 consecutive days initially and twice per week thereafter, for 48-weeks.
  Interventions: Drug: Abatacept (CTLA4-Ig) and nasal placebo (0.9% sodium chloride)

INTERVENTIONS:
Drug: Abatacept (CTLA4-Ig) and nasal insulin (Humulin R®) — Abatacept injected subcutaneously once per week and nasal insulin inhaled for 10 consecutive days initially and twice per week thereafter
  Other Names: Abatacept and nasal insulin
  Arms: Abatacept and nasal insulin
Drug: Abatacept (CTLA4-Ig) and nasal placebo (0.9% sodium chloride) — Abatacept injected subcutaneously once per week and nasal placebo inhaled for 10 consecutive days initially and twice per week thereafter
  Other Names: Abatacept and nasal placebo
  Arms: Abatacept and nasal placebo

SUMMARY:
The goal of this clinical trial is to test whether the combination of two safe immune therapies called abatacept and nasal insulin can preserve pancreas function in recently-diagnosed type 1 diabetes. When type 1 diabetes is first diagnosed, the pancreas is still able to make small amounts of insulin, which helps control glucose levels. Preserving pancreas function can make glucose control easier and reduce the need to use injected insulin.

Participants will be asked to inject abatacept under their skin once per week and inhale nasal insulin or nasal placebo using a spray for 10 consecutive days initially and twice per week thereafter. The treatment period is for 48 weeks, with another 48-week follow-up period.

DETAILED DESCRIPTION:
Type 1 diabetes is caused by an immune attack on insulin-producing beta cells of the pancreas that impairs their ability to make insulin to control blood glucose levels. When diabetes is diagnosed, the pancreas is usually still able to make some insulin, but not enough to meet the body's needs. Over time, continued immune attack further decreases insulin production until after one to two years it is very low or undetectable. When type 1 diabetes is diagnosed, treatments that stop the immune attack may preserve residual beta-cell function. This decreases the requirement for injected insulin and improves glucose control. However, so far, immune therapies have not been shown to prevent ongoing loss of beta-cell function. In this clinical trial, two safe immune therapies called abatacept and nasal insulin will be used together to test if the combination can better preserve the function of beta cells to make insulin after diagnosis. If this occurs, it will be relatively simple to develop this treatment for routine use in recently-diagnosed people and to test whether it prevents high-risk individuals progressing to need insulin injections. This trial will also provide research samples to improve our understanding of how type 1 diabetes develops and how abatacept and nasal insulin might affect this process. The new knowledge created from studying these samples will improve our ability to use abatacept and nasal insulin to preserve pancreas function in type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 21 years and weight at least 20kg at Visit 1
* Diabetes mellitus diagnosed according to ADA criteria (53) within 100 days of Visit 2
* Presence of at least one antibody against insulin (if <10 days since starting insulin therapy), GAD, IA2 or ZnT8
* Random C-peptide >0.3nmol/l, measured by a NATA-accredited pathology laboratory within 2 weeks of Visit 2
* Willing to use CGM for the duration of the study
* Demonstrated ability to record home glucose measurements and insulin doses, as judged by the study doctor
* Willing to forego other forms of experimental treatment during the study
* Fully vaccinated against Covid-19, as recommended by the Australian Technical Advisory Group on Immunisation
* Up to date with other vaccinations recommended by the Australian Technical Advisory Group on Immunisation
* Willing to postpone any live vaccine immunisations for 3 months after treatment

Exclusion Criteria:

* Clinical or laboratory evidence of active infection other than localised skin infection, including viral hepatitis, EBV, CMV or tuberculosis
* Immunodeficiency or chronic use of immunosuppressive drugs other than topical or inhaled glucocorticoid
* Vaccination with live or dead virus within 4 weeks of Visit 2
* History of malignancy
* Pregnant or lactating, or of child-bearing potential not using an effective method of contraception
* Any pathology of the nasal passages that would preclude safe application of the nasal spray
* Any condition that would interfere with study conduct or participant safety

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Beta-cell function at 48 weeks | 0 weeks - 48 weeks
  Change in average C-peptide concentration during a 2-hour mixed meal challenge

SECONDARY OUTCOMES:
Beta-cell function at 24, 72 and 96 weeks | 0, 24, 72 and 96 weeks
  Change in average C-peptide concentration during a 2-hour mixed meal challenge
Glucose regulation | 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72 and 96 weeks
  Proportion of time in the range 3.9-10mmol/l, time below 3.9mmol/l and glucose %CV measured by continuous glucose monitoring (CGM)
Estimated C-peptide concentration | -2, 24, 48, 72 and 96 weeks
  Average C-peptide concentration estimated from fasting glucose, C-peptide, HbA1c, body mass index, disease duration and insulin dose
Frequency of hypoglycemic events | 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60, 72 and 96 weeks
  Frequency of glucose readings <3.0mmol/l, determined by CGM and correcting for CGM wear time
Hemoglobin A1c levels | 0, 12, 24, 36, 48, 60, 72 and 96 weeks
  Change in HbA1c levels
Insulin use | Every 4 weeks for 96 weeks
  Daily insulin dose at all visits
Weight, body mass index and sitting blood pressure | 0, 12, 24, 48, 60, 72 and 96 weeks
  Change in weight, body mass index and blood pressure
Diabetes antibody levels | -2, 0, 4, 12, 24, 48, 60, 72 and 96 weeks
  Insulin, GAD, IA2 and ZnT8 autoantibody concentrations
Quality of life assessment | -2, 0, 24, 48, 72 and 96 weeks
  Assessed by questionnaire
Adverse events | All visits for 96 weeks
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John Wentworth, Principal Investigator — Melbourne Health
Locations (6):
- Australia (6):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - The Royal Melbourne Hospital, Parkville, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to clinical trial — https://atic.svi.edu.au/clinical-trials/